CLINICAL TRIAL: NCT05317650
Title: Effects Multi-Gravitational Suspension-Based Therapy on Posture, Physical Fitness, Quality of Life, Depression, and Sleep Quality in Women Without Regular Exercise Habits
Brief Title: Effects Multi-Gravitational Suspension-Based Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Aybuke Ersin, Head of Physiotherapy and Rehabilitation Department, Atlas University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/128
Record Dates: First submitted 2022-03-02; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Exercise
Keywords: woman; exercise; posture; physical fitness; quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group, no exercise was performed, and the measurements were repeated at the end of 4 weeks.
- M-Gravity group (Experimental): Intervention group performed the exercise with the M-Gravity, 2 sessions per week, for 4 weeks, at the Outpatient Clinic of Department of Physical Therapy, Baskent University, one session for 60 minutes.
  Interventions: Other: Multi-gravitational suspension-based therapy (M-Gravity)

INTERVENTIONS:
Other: Multi-gravitational suspension-based therapy (M-Gravity) — Multi-gravitational suspension-based therapy (M-Gravity) is a comprehensive discipline based on the principles of non-gravity, which serves to increase the quality of life and holistic health of the individual with the rehabilitation content of non-pressure inversion therapy.
  Arms: M-Gravity group

SUMMARY:
Background: Multi-gravitational suspension-based therapy (M-Gravity) is a comprehensive discipline based on the principles of non-gravity, which serves to increase the quality of life and holistic health of the individual with the rehabilitation content of non-pressure inversion therapy.

Aims: To examine the effects of M-Gravity exercise on posture, physical fitness, quality of life, depression, and sleep quality in women without regular exercise habits.

Methods: This study was designed as a non-randomized controlled trial. This study included 20 women without regular exercise habits, who participated in the exercise with M-Gravity and 20 women who did not participate in any exercise program, a total of 40 participants. In this study, the investigators planned to evaluate the effects of M-Gravity on women without regular exercise habits. The following outcomes were measured: posture with the New York Posture Assessment Method, the flexibility of the hamstring and pectoral muscles, time is taken to stay in the plank position, depression levels with the Beck Depression Inventory scale, sleep quality is performed with the Pittsburgh Sleep Quality Index, and the Nottingham Health Profile (NHP) questionnaire to measure the perceived health levels of the subjects. The measurement of the contraction force of the deep lumbar muscles is performed with the Stabilizer Pressure Biofeedback (Chattanooga Stabilizer). Two evaluations were made before and after 4 weeks of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women

Exclusion Criteria:

* Individuals with a physical, cardiac, or neurological disease that may interfere with our practices and assessments
* Pregnancy and post-natal individuals
* Individuals with scoliosis of 20 degrees or more
* Glaucoma
* Recent surgery (3-6 months waiting period according to surgery)
* Hypertension, exercise in the head-down position can cause an increase in blood pressure and a hypertensive crisis
* Impaired cerebral circulation
* Botox treatment in the last 6 hours
* Spinal fractures
* Severe osteoporosis
* Sequestered disc herniation
* Spinal tumors
* Inflammatory conditions of the spine
* Head injuries
* Previous myocardial infarction
* Vertigo

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
New York Posture Assessment Method | 4 weeks
  The posture of the subjects participating in the study was evaluated with the New York Posture Assessment Method (NYPDY). In this evaluation system, postural changes that may occur in 13 different parts of the body were monitored and scored. Accordingly, five (5) points were given if the person's posture was correct, three (3) points if moderately impaired, and one (1) point if severely impaired. The total score obtained as a result of the test is a maximum of 65 and a minimum of 13. Standard evaluation criteria developed for this test were defined as "very good" if the total score is >=45, "good" if the score is 40-44, "moderate" if the score is 30-39, "fair" if the score is 20-29, and "poor" if the score is <=19
Pittsburgh Sleep Quality Index | 4 weeks
  The Pittsburgh Sleep Quality Index, includes 19 questions and consists of seven items evaluating subjective sleep quality, sleep delay, sleep duration, sleep efficiency, sleep disturbance, use of sleeping pills, and impairment in daytime work. The response of each is scored between 0-3 according to symptom frequency. Scoring; 0 if it has never happened during the past month, 1 if it is less than once a week, 2 if it is once or twice a week, and 3 if it is three or more times a week. The sleep quality assessment asked in the questionnaire is; It is scored as 0 very good, 1 fairly good, 2 very badly, and 3 very badly. The obtained global score ranges from 0 to 21, and high values indicate poor sleep quality and high level of sleep disturbance. A global score of 5 or above indicates that the quality of sleep is clinically significantly worse.
Nottingham Health Profile | 4 weeks
  The 'Nottingham Health Profile is a general quality of life questionnaire that measures the perceived health problems of the person and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), emotional reactions (9 items). Each sub-parameter is scored between 0-100. 0 indicates best health, 100 indicates worst health.
Stabilizer Pressure Biofeedback | 4 weeks
  The measurement of the contraction force of the deep lumbar muscles is performed with the "Stabilizer Pressure Biofeedback" (Chattanooga Stabilizer). Before the test, each patient is taught how to tighten the Transversus Abdominous with the corset method in the supine and quadrupedal position. Subjects will be placed face down on an inflated pillow attached to a manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Aybüke Ersin, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No